CLINICAL TRIAL: NCT00220545
Title: A Prospective Randomized Controlled Trial to Compare Laparoscopic Ovarian Diathermy With Clomiphene Citrate as a First Line Treatment of Anovulatory Infertility in Patients With Polycystic Ovarian Syndrome
Brief Title: Comparison Between Laparoscopic Ovarian Diathermy and Clomiphene Citrate in Women With Anovulatory PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH5735 01/173
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovarY; Laparoscopic ovarian diathermy; Induction of ovulation; Clomiphene citrate
MeSH Terms: conditions — Polycystic Ovary Syndrome

INTERVENTIONS:
Procedure: Laparoscopic ovarian diathermy

SUMMARY:
Laparoscopic ovarian diathermy (LOD) is currently offered to infertile women with polycystic ovarian syndrome (PCOS) who fail to conceive on clomiphene citrate (CC). However, using LOD before CC may result in a better reproductive outcome since LOD may reduce risks associated with CC such as miscarriages and multiple pregnancies. The aim of the study is to evaluate the effectiveness of LOD and its potential value in improving the success rates in infertile women with PCOS. This study will recruit 72 women with PCOS suffering from infertility due to lack of ovulation from the infertility clinic. After initial assessment, patients will be given explanation about the study and will receive an information leaflet. They will then be randomized into two groups: Group1 (36 patients) will receive CC as per infertility clinic protocol to induce ovulation for up to 6 months. Group 2 (36 patients) will undergo laparoscopic ovarian diathermy under general anaesthetic. Blood samples will be taken from both groups before any treatment, shortly after treatment and at 3 and 6 months after treatment to measure various hormones. Patients will be contacted every month after treatment for follow up. The reproductive outcomes particularly the pregnancy and livebirth rates will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19 - 39
2. BMI < 32
3. Anovulatory Infertility > 1 year
4. Diagnostic criteria for
5. No previous treatment for induction of ovulation
6. Normal semen analysis of partner
7. Proven patency of at least one Fallopian tube

Exclusion Criteria:

1. Inability to give informed consent
2. Contraindication to CC
3. Contraindication to general anaesthetic or laparoscopy

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2002-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Pregnancy rates

SECONDARY OUTCOMES:
Ovulation, Pregnancy outcome (especially miscarriage), Menstrual pattern, Endocrine changes, Side effects / complications rate

CONTACTS AND LOCATIONS:
Overall Officials: Saad AK Amer, MD, Principal Investigator — University of Sheffield
Locations (1):
- Jessop Wing, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Amer SA, Li TC, Metwally M, Emarh M, Ledger WL. Randomized controlled trial comparing laparoscopic ovarian diathermy with clomiphene citrate as a first-line method of ovulation induction in women with polycystic ovary syndrome. Hum Reprod. 2009 Jan;24(1):219-25. doi: 10.1093/humrep/den325. Epub 2008 Sep 14. PMID 18794162